CLINICAL TRIAL: NCT04337398
Title: Feasibility, Adherence and Effects of Two Exercise-based Interventions in Adults With Severe Mental Illness. The PsychiActive Project 2.0
Brief Title: Exercise in Severe Mental Illness. The PsychiActive Project 2.0
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Pablo de Olavide (Other)
Responsible Party: Principal Investigator, Alvaro López Moral, MSc Sport Sciences, Universidad Pablo de Olavide
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTS948AFS20
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Exercise Therapy; Severe Mental Illness
Keywords: Exercise; Severe Mental Illness; Adherence; Wearables; Activity Trackers; Exergames
MeSH Terms: conditions — Mental Disorders; Motor Activity | interventions — Exercise; Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearables (Experimental): Adults with several mental illness
  Interventions: Behavioral: Exercise training for 12 weeks (wearables)
- Wearables and exergames (Experimental): Adults with several mental illness
  Interventions: Behavioral: Exercise training for 12 weeks (wearables and exergames)

INTERVENTIONS:
Behavioral: Exercise training for 12 weeks (wearables) — Activity trackers with adaptive weekly step goals, weekly walking groups and coaching.
  Other Names: Xiaomi MiBand4
  Arms: Wearables
Behavioral: Exercise training for 12 weeks (wearables and exergames) — Activity trackers with adaptive weekly step goals, weekly walking groups, coaching and exercise programme based on exergames (aerobic, resistance and stretching training three weekly group sessions).
  Other Names: Xiaomi MiBand4 and Xbox 360 Kinect
  Arms: Wearables and exergames

SUMMARY:
The purpose of this randomized controlled trial is to study the feasibility, adherence and effects of two exercise interventions on body weight, body composition, anthropometric and fasting blood measures, physical fitness, quality of life, and lifestyle habits in patients with severe mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psychiatric disorder (ICD-10).
* Stabilized antipsychotic medication during the last month.

Exclusion Criteria:

* Clinical instability.
* Substance abuse.
* Comorbidities contraindicating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported sedentary behavior | 12 weeks
  In hours per week. Using the Sedentary Behaviour Questionnaire. It asks about amount of time spent doing 11 sedentary behaviours of a usual weekday and weekend day. Time in hours of each behaviour were summed separately for weekdays and weekend days, and time for an average day was calculated as (weekday hours ×5 +weekend day hours × 2)/7. Higher values represent a higher level of sedentary behavior.
Self-reported physical activity | 12 weeks
  In metabolic equivalent minutes per week. Using the Simple Physical Activity Questionnaire. Higher values represent a higher level of physical activity.
Behavioral Regulation in Exercise | 12 weeks
  Using the Behavioral Regulation in Exercise Questionnaire. It consists of 24 items1 with a five-point Likert scale, which varied between 1 ("Strongly Disagree") and 4 ("Strongly Agree"). The items were grouped posteriorly into six factors (with four items each). Higher values represent a higher level of motivational continuum of self-determination theory.
Adherence | 12 weeks
  In percent. Adherence will be evaluated by the percentage of attendance with respect to the total number of minutes of intervention.
Dropout | 12 weeks
  In percent. Dropout will be study by the percent drop relative to the total subjects began intervention.
Body weight | 12 weeks
  In kilograms. Using the InBody 770 Body Composition Analyzer (Biospace Ltd, Seoul, Korea)
Fat mass | 12 weeks
  In kilograms. Using the InBody 770 Body Composition Analyzer (Biospace Ltd, Seoul, Korea)
Lean mass | 12 weeks
  In kilograms. Using the InBody 770 Body Composition Analyzer (Biospace Ltd, Seoul, Korea)
Waist circumference | 12 weeks
  In millimeters. Using a measuring tape (Harpenden Anthropometric Tape; Holtain, Dyfed, UK) placed at the midpoint between the last rib and the iliac crest
Hip circumference | 12 weeks
  In millimeters. Using a measuring tape (Harpenden Anthropometric Tape; Holtain, Dyfed, UK) placed atthe maximum width over the greater trochanters
Health status | 12 weeks
  Using the Short Form 36-Item Health Survey questionnaire version 2. Examines eight domains of physical (physical functioning, physical role, body pain, and general health) and mental health status (vitality, social functioning, emotional role, and mental health). The four physical-domains are summarized into a physical component score, and the four mental-domains constitute a mental component score. Scores range from 0 to 100 points, with higher scores indicating better health status.
Quality of Life | 12 weeks
  Using the European Quality of Life-5 Dimensions Questionnaire.The descriptive system contains five dimensions of health (mobility, personal care, daily activities, pain / discomfort and anxiety / depression) and each of them has three levels of severity (no problems, some moderate or severe problems and problems). Scores range from 0 to 1 point, with higher scores indicating better quality of life.
Self-Reported Physical Fitness | 12 weeks
  Using "The International Fitness Scale" (IFIS) questionnaire. The IFIS consists of a Likert-type scale (range 1-5) with five response options (very poor, poor, average, good, and very good) about perceived overall fitness, and its main components are cardiorespiratory fitness, muscular strength, speed-agility, and flexibility. Higher scores indicating better physical fitness.

SECONDARY OUTCOMES:
Lower body strength | 12 weeks
  In number of full stands. Using the 30-second chair stand test
Upper body strength | 12 weeks
  In number of bicep curls. Using the 30-second arm curl test.
Handgrip strength | 12 weeks
  In kilograms. Using a dynamometer (TKK 5401 Grip-D, Takey, Tokyo, Japan)
Cardiorespiratory fitness | 12 weeks
  In meters. Using the 6-min walk test.
Lower body flexibility | 12 weeks
  In centimeters. Using the chair sit-and-reach test
Upper body flexibility | 12 weeks
  In centimeters. Using the back scratch test
Mood | 12 weeks
  Using the Scale for Mood Assessment. This questionnaire valuates four moods through 16 items divided into four categories: sadness-depression, anxiety, anger/hostility and happiness. Item scores are evaluated with the Likert scales ranging from 0 to 10, higher values represent a higher level of this mood.
Psychopathological symptoms | 12 weeks
  Using the Brief Symptom Inventory-18 questionnaire. Score range from 0 to 72 points. Higher values represent a higher psychopathological severity.
Smoking | 12 weeks
  Using the Fagerström nicotine dependence questionnaire. Score range from 0 to 10 points. Higher values represent a higher nicotine dependece.
Blood glucose | 12 weeks
  In milligram per deciliter. Collected in the morning after an overnight fast
Blood cholesterol | 12 weeks
  In milligram per deciliter. Collected in the morning after an overnight fast
Blood triglyceride | 12 weeks
  In milligram per deciliter. Collected in the morning after an overnight fast

CONTACTS AND LOCATIONS:
Overall Officials: Diego Munguía-Izquierdo, PhD, Principal Investigator — Universidad Pablo de Olavide
Locations (1):
- Álvaro López Moral, Seville, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No